CLINICAL TRIAL: NCT07268534
Title: Biologics in Folliculitis Decalvans : an Adaptative Trial Research
Acronym: BOOSTERS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP230831; 2024-514848-88-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-04; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Folliculitis Decalvans (FD)
Keywords: Folliculitis Decalvans; FD; alopecia; TNFa inhibitor; IL12 inhibitor; IL23 inhibitor; JAK1 inhibitor; JAK2 inhibitor
MeSH Terms: conditions — Alopecia | interventions — Adalimumab; Ustekinumab; baricitinib

STUDY DESIGN:
Intervention Model Description: This is a national multicenter, randomized, not controlled single-blind, phase II clinical study.The study will be considered in a general Bayesian framework. The design is not conceived for between-group comparisons but to potentially individualize promising treatment allowing early stop of treatment based on unacceptable posterior probability of success.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational medicinal product 1 (Experimental): 1) Adalimumab = TNFa inhibitor
  Interventions: Drug: Adalimumab
- Investigational medicinal product 2 (Experimental): 2) Ustekinumab = IL12 and 23 inhibitor
  Interventions: Drug: Ustekinumab
- Investigational medicinal product 3 (Experimental): 3) Baricitinib = inhibitor JAK 1 and JAK 2
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Adalimumab — For a 6-month duration
  Arms: Investigational medicinal product 1
Drug: Ustekinumab — For a 6-month duration
  Arms: Investigational medicinal product 2
Drug: Baricitinib — For a 6-month duration
  Arms: Investigational medicinal product 3

SUMMARY:
FD (which was in the past named Quinquaud folliculitis) is a rare disease defined by a chronic, neutrophilic folliculitis of the scalp, leading to scarring alopecia. During the flares, scabs and pustules, sometimes very extensive and painful, induce definitive alopecia with quality of life is considerably impaired. Pathophysiology remains unclear although the cutaneous microbiota with a rupture of the epidermal barrier, leading to pathogen invasion, most often Staphylococcus aureus (SA), has been involved.It explains why first-line treatment of FD is antibiotics, i.e., oral tetracycline/doxycycline (combined with topical antibiotics) for 3 months at least. Second-line treatment includes an association of antibiotics, e.g., rifampicin-clindamycin for 10-12 weeks or, in case of contraindication or unavaibility of one or both of these drugs, other antibiotics listed.

Short-term efficacy rate of antibiotics is around 50-60%, but unfortunately, recurrences/relapses are occurring 5 to 7 months on average after stopping antibiotics, requiring their reintroduction/long-term use and potentially less efficacy/ecological harms. So far, FD is a non-curable disease for which inflammatory pathways involving several cytokines as TNF, IL1β, IL8, TGFβ, IL12 and 23, could also play a role.

DETAILED DESCRIPTION:
Folliculitis Decalvans (FD) is a rare disease defined by a chronic, neutrophilic folliculitis of the scalp, leading to scarring alopecia. During the flares, scabs and pustules, sometimes very extensive and painful, induce the definitive alopecia. As expected, quality of life is heavily impaired. Pathophysiology remains unclear although the microbiota with a rupture of the epidermal barrier, leading to pathogen invasion, most often Staphylococcus aureus (SA), has been involved. It explains why first-line treatment of FD is antibiotics, i.e., oral tetracycline / doxycycline (combined with topical antibiotics) for 3 months at least. Second-line treatment includes an association of antibiotics, e.g., rifampicin-clindamycin for 10-12 weeks.

Short-term efficacy level of antibiotics is around 50-60% but unfortunately, recurrences/relapses are occurring 5 to 7 months after stopping antibiotics on average, requiring their reintroduction/long-term use and potentially less efficacy. So far, FD is a non-curable disease for which inflammatory pathways involving several cytokines as TNF, IL1β, IL8, TGFβ, IL12, IL 23, could also play a role. The similarity of FD with hidradenitis suppurativa (HS) suggests a double approach based on antibiotics and immunomodulatory targeted drugs. Only short series have been reported in attempting to control the inflammatory response by biologic agents, including anti-TNF, anti-IL12 and IL23, JAK inhibitors. Although several cures of antibiotics could be delivered lifelong, it may impair the microbiota at the individual and populational levels with known (and possibly still unknown) ecological consequences. With regards to limited available treatment, potential harms of antibiotics, and absence of therapeutic strategy, any new treatment able to control signs and symptoms of flare of FD in patients previously treated by 2 lines of antibiotics - so called difficult-to- treat patients - could be used in a forthcoming strategy.

We hypothesized that targeted therapies as biologics could control a flare of FD in difficult-to-treat patients with a relevant response. With regards to the literature, this approach would allow a new clue in the management of FD.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18-year-old and < 65-year-old
* Presenting with FD confirmed in all cases by at least one compatible histopathology (present or past)
* All patients should have a basal FD-IGA score at 3 or 4 and should have received in the previous 2 years at least two lines of antibiotics (first line : at least 3 months doxy/lymecycline (doxycycline 200 mg/day or at least 2 weeks, then 100 mg/day in the following weeks, or lymecycline 300 mg/day for at least 2 weeks, then 150 mg/day in the following weeks) ; second line : Rifampicin/clindamycin 10 weeks (classic regimen for FD) or, in case of contraindication or unaivailability of one or both of these drugs, other antibiotics prescribed for at least 3 weeks alone or in combination (list of antibiotics).
* Normal chest x-ray less than 3 months old on the day of inclusion
* Individuals affiliated to a social security regimen
* Individuals able to understand and express himself/herself in French
* Individuals able to participate and to follow up during the study period
* Written informed consent from the patient

The diagnosis of Folliculitis Decalvans must have been validated collectively as part of care with at least one FD expert.

Exclusion Criteria:

* Patients with a history of cardiac ischaemia
* Moderate to severe heart failure (NYHA classes III/IV)

As the whole treatment duration will only be 6 months, the risk of baricitinib-related SAEs will be minimized according to the recent PRAC from the EMA by excluding:

* Patients at increased risk of major cardio-vascular problem,
* Patients heavy smokers (25 cig/day),
* Current or past history of malignancy, with the exception of non-melanoma skin cancer excised and cured more than five years before baseline, per investigator assessment.

  * Morbid obesity: BMI > 40
  * Individuals with known positive HIV tests and any immunosuppressive condition or drugs.
  * Hypersensitivity to the active substance or to any of the excipients: Adalimumab, Ustekinumab, Baricitinib (see SmPC)
  * Patient who has already received one of the treatments evaluated (Adalimumab, Ustekinumab, Baricitinib).
  * Patient with renal insufficiency (creatinine clearance < 60 mL/min)
  * Coexisting inflammatory facial dermatosis such as acne fulminans, hidradenitis suppurativa
  * Active tuberculosis or other severe infections such as sepsis and opportunistic infections
  * Women who are pregnant or are breast-feeding, or are of childbearing age who have not used or do not plan to use acceptable birth control measures
  * Individuals under a measure of legal protection or unable to consent
  * Participation in another interventional study involving human participants or in the exclusion period at the end of a previous study involving human participants, if applicable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
The primary end point is an IGA score (FD-IGA) which will be assessed by a blinded assessor. Success will be defined by at least a decrease of 2 points of the FD-IGA at 6 month | At 6 month

SECONDARY OUTCOMES:
Pain evaluated by Visual analogue Scale (VAS) at randomization, 3, 6 and 12 months | at 3, 6 and 12 months
Pain change from randomization, at 3, 6 and 12 months | at 3, 6 and 12 months
Pruritus evaluated by Worst Itch Numeric Rating Scale (WI-NRS) at randomization, 3, 6 and 12 months | at 3, 6 and 12 months
Quality of life evaluated by Dermatology life quality index (DLQI) at randomization, 3, 6 and 12 months | at 3, 6 and 12 months
Time to first relapse during the study period | during the study period
Measure of FD-IGA score in the population of patients receiving the antibiotic rescue (at the onset of the rescue) | at the onset of the rescue
Measure of FD-IGA score (blinded assessor) at 12 months | at 12 months
Tolerance of drugs | during the study period

IPD SHARING:
Plan to Share IPD: No